CLINICAL TRIAL: NCT00640250
Title: Clinical Evaluation of T.R.U.E. TEST® Panel 3.2 Allergens: Bronopol and Disperse Blue 106 Dose Response Study
Brief Title: Clinical Evaluation of T.R.U.E. TEST® Panel 3.2 Allergens: Dose Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allerderm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Mekos 07 2P3.2 201; 2007-007130-19 (EudraCT Number); WIRB Pr. No.: 20072233 (Other: Western Institutional Review Board)
Record Dates: First submitted 2008-03-03; First posted 2008-03-21 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Contact Dermatitis
Keywords: Dermatitis, Contact, Bronopol, Disperse Blue 106
MeSH Terms: conditions — Dermatitis, Contact; Dermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sensitives (Experimental): Subjects with a clinical history and positive patch test (current or previous) to either Disperse Blue 106 or Bronopol. Subjects must otherwise be healthy and fulfill entry criteria.
  Interventions: Biological: T.R.U.E. TEST® Skin Patch Test: Dose Response Allergens

INTERVENTIONS:
Biological: T.R.U.E. TEST® Skin Patch Test: Dose Response Allergens — Disperse blue 106 in PVP, 0.15 mg/cm2 Disperse blue 106 in PVP, 0.050 mg/cm2 Disperse blue 106 in PVP, 0.017 mg/cm2 PVP Negative Control Bronopol in PVP, 0.75 mg/cm2 Bronopol in PVP, 0.50 mg/cm2 Bronopol in PVP, 0.25 mg/cm2 Bronopol in PVP, 0.125 mg/cm2
  Test patches, with allergens, are placed at day one and removed 48 hours later. The duration of the study lasts 21 days. However, the subject is only exposed to the study allergens for 48 hours.
  Other Names: T.R.U.E. TEST® Skin Patch Test: Panel 3.2

SUMMARY:
We propose a prospective, multi-center, double-blind, randomized study comparing the diagnostic performance (primary) and safety (secondary) of 3 concentrations of Disperse blue 106 and 4 concentrations of Bronopol in 40 adult subjects (20 subjects per allergen) with a clinical history of contact dermatitis and a positive patch test (current or previous) to the corresponding reference petrolatum allergen ("sensitives").

DETAILED DESCRIPTION:
Primary endpoint:

To evaluate the diagnostic performance of Disperse blue 106 and Bronopol T.R.U.E. Test allergens in 20 adult subjects per allergen with a clinical history of contact dermatitis and a positive patch test to the respective reference allergen. Evaluations will include:

* Determination of the lowest concentration eliciting positive skin reactions (+1 or +2) in 70-90% of sensitive subjects.
* Frequency of positive, negative, doubtful and irritant reactions for each allergen and tested concentration.
* Concordance/discordance as compared to the corresponding reference petrolatum allergen.

Secondary endpoint:

To evaluate the safety of Disperse blue 106 and Bronopol T.R.U.E. Test allergens in 20 adult subjects per allergen with a clinical history of contact dermatitis and a positive patch test to the respective reference allergen. Evaluations will include:

* The frequency of tape-induced irritation at the test site, incomplete panel adhesion, and subject-reported sensations of itching or burning.
* The frequency and characterization of adverse events and serious adverse events.
* The frequency and characterization of late and/or persistent reactions.

ELIGIBILITY:
Inclusion Criteria:

* Current or previous symptoms and/or history consistent with allergic contact dermatitis, and positive patch test (within the past 5 years) to Bronopol OR Current or previous symptoms and/or history consistent with allergic contact dermatitis, and a positive patch test (within the past 5 years) to Disperse blue 106 or Disperse blue 106/124 allergen mix.
* All subjects must be adults (18 years of age or older) and otherwise in good health.
* Premenopausal female subjects must consent to a urine pregnancy test; results must be negative for study inclusion.
* Informed consent must be signed and understood by each subject, and consistent with all institutional, local and national regulations.

Exclusion Criteria:

* Subjects unable to meet inclusion requirements.
* Women who are breastfeeding or pregnant.
* Topical treatment during the last 7 days with corticosteroids or other immunosuppressive agents on or near the test area.
* Systemic treatment during the last 7 days with corticosteroids (equivalent to > 10 mg prednisone) or other immunosuppressive agents.
* Treatment with ultraviolet (UV) light (including tanning) during the previous 3 weeks.
* Acute dermatitis outbreak or dermatitis on or near the test area on the back.
* Subjects unable to comply with patch test study requirements including multiple return visits and activity restrictions (e.g., protecting test panels from excess moisture due to showering or vigorous activity).
* Subject participation in clinical trials of investigational drugs, treatments or devices other than T.R.U.E. Test during this study or 3 weeks prior to inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evy Paulsen, M.D., Ph.D, Principal Investigator — Odense University Hospital; Joseph Fowler, MD, Principal Investigator — Dermatology Specialists PSC
Locations (2):
- Dermatology Specialists PSC, Louisville, Kentucky, United States
- Odense University Hospital, Odense C, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: 16 June 2008 through 7 April 2009. This study was conducted at two investigational sites located in Denmark (E Paulsen) and the United States (J Fowler).
Pre-assignment Details: There were no significant events or approaches which caused enrolled participants to be excluded from the trial before assignment to a group.
Period: Overall Study
Arm/Group | Sensitives
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The analysis included all enrolled subjects but it should be noted that subject 5-D220 was not sensitive to either allergen and thus was not included in either population of sensitive subjects; the subject was included in the population of all enrolled subjects.
Arm/Group | Sensitives
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 27
  Denmark | 21

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Performance: Optimal Test Allergen Concentration
Description: Lowest concentration eliciting 1+ or 2+ positive reactions in 70-90% of subjects
Time Frame: Visits 3-5: 3-21 days after application
Population: Percentage is based on subjects sensitive to each allergen. Results from one subject not included due to no past history of positive patch test.
Measure: Number; unit: percentage of participants
Groups:
- Disperse Blue 0.017 mg/cm2; Disperse Blue 0.050 mg/cm2; Disperse Blue 0.150 mg/cm2; Bronopol 0.125 mg/cm2; Bronopol 0.250 mg/cm2; Bronopol 0.500 mg/cm2; Bronopol 0.750 mg/cm2: Percentage of positive test responses
Arm/Group | Disperse Blue 0.017 mg/cm2 | Disperse Blue 0.050 mg/cm2 | Disperse Blue 0.150 mg/cm2 | Bronopol 0.125 mg/cm2 | Bronopol 0.250 mg/cm2 | Bronopol 0.500 mg/cm2 | Bronopol 0.750 mg/cm2
Number analyzed (Participants) | 21 | 21 | 21 | 26 | 26 | 26 | 26
percentage of participants | 38.1 | 47.6 | 52.4 | 30.8 | 23.1 | 46.2 | 61.5

2. Primary Outcome: Frequency of Positive, Negative, Doubtful and Irritant Reactions for Each Allergen and Concentration
Description: Percentage (including confidence intervals) of subjects who elicited positive, negative, doubtful and irritant reactions to disperse blue at visit 3- all subjects
Time Frame: Visit 3: 3 days after application
Population: All subjects
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Disperse Blue 0.017 mg/cm2 Positive Reactions; Disperse Blue 0.050 mg/cm2 Positive Reactions; Disperse Blue 0.150 mg/cm2 Positive Reactions; Negative Control Positive Reactions: Percentage of subjects who exhibited positive reactions at visit 3
- Disperse Blue 0.017 Negative Reactions; Disperse Blue 0.050 mg/cm2 Negative Reactions; Disperse Blue 0.150 mg/cm2 Negative Reactions; Negative Control Negative Reactions: Percentage of subjects who exhibited negative reactions at visit 3
- Disperse Blue 0.017 mg/cm2 Irritant Reactions; Disperse Blue 0.050 mg/cm2 Irritant Reactions; Disperse Blue 0.150 mg/cm2 Irritant Reactions; Negative Control Irritant Reactions: Percentage of subjects who exhibited irritant reactions at visit 3
- Disperse Blue 0.017 mg/cm2 Doubtful Reactions; Disperse Blue 0.050 mg/cm2 Doubtful Reactions; Disperse Blue 0.150 mg/cm2 Doubtful Reactions; Negative Control Doubtful Reactions: Percentage of subjects who exhibited doubtful reactions at visit 3
Arm/Group | Disperse Blue 0.017 mg/cm2 Positive Reactions | Disperse Blue 0.050 mg/cm2 Positive Reactions | Disperse Blue 0.150 mg/cm2 Positive Reactions | Negative Control Positive Reactions | Disperse Blue 0.017 Negative Reactions | Disperse Blue 0.050 mg/cm2 Negative Reactions | Disperse Blue 0.150 mg/cm2 Negative Reactions | Negative Control Negative Reactions | Disperse Blue 0.017 mg/cm2 Irritant Reactions | Disperse Blue 0.050 mg/cm2 Irritant Reactions | Disperse Blue 0.150 mg/cm2 Irritant Reactions | Negative Control Irritant Reactions | Disperse Blue 0.017 mg/cm2 Doubtful Reactions | Disperse Blue 0.050 mg/cm2 Doubtful Reactions | Disperse Blue 0.150 mg/cm2 Doubtful Reactions | Negative Control Doubtful Reactions
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48
percentage of participants | 16.7 [7.5 to 30.2] | 18.8 [8.9 to 32.6] | 25.0 [13.6 to 39.6] | 2.1 [0.1 to 11.1] | 75.0 [60.4 to 86.4] | 77.1 [62.7 to 88.0] | 72.9 [58.2 to 84.7] | 91.7 [80.0 to 97.7] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.4] | 8.3 [2.3 to 20.0] | 4.2 [0.5 to 14.3] | 2.1 [0.1 to 11.1] | 6.3 [1.3 to 17.2]

3. Primary Outcome: Frequency of Positive, Negative, Doubtful and Irritant Reactions for Each Allergen and Concentration
Description: Percent (including confidence intervals) of subjects who elicited positive, negative, doubtful and irritant reactions to disperse blue at visit 4- all subjects
Time Frame: Visit 4: 7 days after application
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Disperse Blue 0.017 mg/cm2 Positive Reactions; Disperse Blue 0.050 mg/cm2 Positive Reactions; Disperse Blue 0.150 mg/cm2 Positive Reactions; Negative Control Positive Reactions: Percentage of subjects who exhibited positive reactions at visit 4
- Disperse Blue 0.017 Negative Reactions; Disperse Blue 0.050 mg/cm2 Negative Reactions; Disperse Blue 0.150 mg/cm2 Negative Reactions; Negative Control Negative Reactions: Percentage of subjects who exhibited negative reactions at visit 4
- Disperse Blue 0.017 mg/cm2 Irritant Reactions; Disperse Blue 0.050 mg/cm2 Irritant Reactions; Disperse Blue 0.150 mg/cm2 Irritant Reactions; Negative Control Irritant Reactions: Percentage of subjects who exhibited irritant reactions at visit 4
- Disperse Blue 0.017 mg/cm2 Doubtful Reactions; Disperse Blue 0.050 mg/cm2 Doubtful Reactions; Disperse Blue 0.150 mg/cm2 Doubtful Reactions; Negative Control Doubtful Reactions: Percentage of subjects who exhibited doubtful reactions at visit 4
Arm/Group | Disperse Blue 0.017 mg/cm2 Positive Reactions | Disperse Blue 0.050 mg/cm2 Positive Reactions | Disperse Blue 0.150 mg/cm2 Positive Reactions | Negative Control Positive Reactions | Disperse Blue 0.017 Negative Reactions | Disperse Blue 0.050 mg/cm2 Negative Reactions | Disperse Blue 0.150 mg/cm2 Negative Reactions | Negative Control Negative Reactions | Disperse Blue 0.017 mg/cm2 Irritant Reactions | Disperse Blue 0.050 mg/cm2 Irritant Reactions | Disperse Blue 0.150 mg/cm2 Irritant Reactions | Negative Control Irritant Reactions | Disperse Blue 0.017 mg/cm2 Doubtful Reactions | Disperse Blue 0.050 mg/cm2 Doubtful Reactions | Disperse Blue 0.150 mg/cm2 Doubtful Reactions | Negative Control Doubtful Reactions
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48
percentage of participants | 18.8 [8.9 to 32.6] | 18.8 [8.9 to 32.6] | 27.1 [15.3 to 41.8] | 0.0 [0.0 to 7.4] | 75.0 [60.4 to 86.4] | 72.9 [58.2 to 84.7] | 70.8 [55.9 to 83.0] | 97.9 [88.9 to 99.9] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.4] | 6.3 [1.3 to 17.2] | 8.3 [2.3 to 20.0] | 2.1 [0.1 to 11.1] | 2.1 [0.1 to 11.1]

4. Primary Outcome: Frequency of Positive, Negative, Doubtful and Irritant Reactions for Each Allergen and Concentration
Description: Percentage (including confidence intervals) of subjects who exhibited positive, negative, doubtful and irritant reactions to bronopol at visit 3- all subjects
Time Frame: Visit 3: 3 days after application
Population: Data from one subject not included because subject did not have a past positive response to either allergen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Bronopol 0.1 mg/cm2 Positive Reactions; Bronopol 0.250 mg/cm2 Positive Reactions; Bronopol 0.500 mg/cm2 Positive Reactions; Bronopol 0.750 mg/cm2 Positive Reactions: Percentage of subjects who exhibited positive reactions at visit 3
- Bronopol 0.1 Negative Reactions; Bronopol 0.250 mg/cm2 Negative Reactions; Bronopol 0.500 mg/cm2 Negative Reactions; Bronopol 0.750 mg/cm2 Negative Reactions: Percentage of subjects who exhibited negative reactions at visit 3
- Bronopol 0.1 mg/cm2 Irritant Reactions; Bronopol 0.250 mg/cm2 Irritant Reactions; Bronopol 0.500 mg/cm2 Irritant Reactions; Bronopol 0.750 mg/cm2 Irritant Reactions: Percentage of subjects who exhibited irritant reactions at visit 3
- Bronopol 0.1 mg/cm2 Doubtful Reactions; Bronopol 0.250 mg/cm2 Doubtful Reactions; Bronopol 0.500 mg/cm2 Doubtful Reactions; Bronopol 0.750 mg/cm2 Doubtful Reactions: Percentage of subjects who exhibited doubtful reactions at visit 3
Arm/Group | Bronopol 0.1 mg/cm2 Positive Reactions | Bronopol 0.250 mg/cm2 Positive Reactions | Bronopol 0.500 mg/cm2 Positive Reactions | Bronopol 0.750 mg/cm2 Positive Reactions | Bronopol 0.1 Negative Reactions | Bronopol 0.250 mg/cm2 Negative Reactions | Bronopol 0.500 mg/cm2 Negative Reactions | Bronopol 0.750 mg/cm2 Negative Reactions | Bronopol 0.1 mg/cm2 Irritant Reactions | Bronopol 0.250 mg/cm2 Irritant Reactions | Bronopol 0.500 mg/cm2 Irritant Reactions | Bronopol 0.750 mg/cm2 Irritant Reactions | Bronopol 0.1 mg/cm2 Doubtful Reactions | Bronopol 0.250 mg/cm2 Doubtful Reactions | Bronopol 0.500 mg/cm2 Doubtful Reactions | Bronopol 0.750 mg/cm2 Doubtful Reactions
Number analyzed (Participants) | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47
percentage of participants | 14.6 [6.1 to 27.8] | 14.6 [6.1 to 27.8] | 25.0 [13.6 to 39.6] | 45.8 [31.4 to 60.8] | 79.2 [65.0 to 89.5] | 72.9 [58.2 to 84.7] | 58.3 [43.2 to 72.4] | 37.5 [24.0 to 52.6] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 7.4] | 2.1 [0.1 to 11.1] | 0.0 [0.0 to 7.4] | 6.3 [1.3 to 17.2] | 12.5 [4.7 to 25.2] | 14.6 [6.1 to 27.8] | 16.7 [7.5 to 30.2]

5. Primary Outcome: Frequency of Positive, Negative, Doubtful and Irritant Reactions for Each Allergen and Concentration
Description: Percentage (including confidence intervals) of subjects who exhibited positive, negative, doubtful and irritant reactions to bronopol at visit 4- all subjects
Time Frame: Visit 4: 7 days after application
Population: Data from one subject not included because subject did not have past positive response to either allergen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Bronopol 0.125 mg/cm2 Positive Reactions; Bronopol 0.250 mg/cm2 Positive Reactions; Bronopol 0.500 mg/cm2 Positive Reactions; Bronopol 0.750 mg/cm2 Positive Reactions: Percentage of subjects who exhibited positive reactions at visit 4
- Bronopol 0.125 Negative Reactions; Bronopol 0.250 mg/cm2 Negative Reactions; Bronopol 0.500 mg/cm2 Negative Reactions; Bronopol 0.750 mg/cm2 Negative Reactions: Percentage of subjects who exhibited negative reactions at visit 4
- Bronopol 0.125 mg/cm2 Irritant Reactions; Bronopol 0.250 mg/cm2 Irritant Reactions; Bronopol 0.500 mg/cm2 Irritant Reactions; Bronopol 0.750 mg/cm2 Irritant Reactions: Percentage of subjects who exhibited irritant reactions at visit 4
- Bronopol 0.125 mg/cm2 Doubtful Reactions; Bronopol 0.250 mg/cm2 Doubtful Reactions; Bronopol 0.500 mg/cm2 Doubtful Reactions; Bronopol 0.750 mg/cm2 Doubtful Reactions: Percentage of subjects who exhibited doubtful reactions at visit 4
Arm/Group | Bronopol 0.125 mg/cm2 Positive Reactions | Bronopol 0.250 mg/cm2 Positive Reactions | Bronopol 0.500 mg/cm2 Positive Reactions | Bronopol 0.750 mg/cm2 Positive Reactions | Bronopol 0.125 Negative Reactions | Bronopol 0.250 mg/cm2 Negative Reactions | Bronopol 0.500 mg/cm2 Negative Reactions | Bronopol 0.750 mg/cm2 Negative Reactions | Bronopol 0.125 mg/cm2 Irritant Reactions | Bronopol 0.250 mg/cm2 Irritant Reactions | Bronopol 0.500 mg/cm2 Irritant Reactions | Bronopol 0.750 mg/cm2 Irritant Reactions | Bronopol 0.125 mg/cm2 Doubtful Reactions | Bronopol 0.250 mg/cm2 Doubtful Reactions | Bronopol 0.500 mg/cm2 Doubtful Reactions | Bronopol 0.750 mg/cm2 Doubtful Reactions
Number analyzed (Participants) | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47 | 47
percentage of participants | 14.9 [6.2 to 28.3] | 17.0 [7.6 to 30.8] | 21.3 [10.7 to 35.7] | 29.8 [17.3 to 44.9] | 78.7 [64.3 to 89.3] | 74.5 [59.7 to 86.1] | 59.6 [44.3 to 73.6] | 57.4 [42.2 to 71.7] | 0.0 [0.0 to 7.5] | 0.0 [0.0 to 7.5] | 4.3 [0.5 to 14.5] | 8.5 [2.4 to 20.4] | 6.4 [1.3 to 17.5] | 8.5 [2.4 to 20.4] | 14.9 [6.2 to 28.3] | 4.3 [0.5 to 14.5]

6. Primary Outcome: Concordance Between Investigational Allergen and Reference Allergen
Description: Concordance between disperse blue or bronopol and the respective reference petrolatum allergen
Time Frame: Visit 5: 21 days after patch application
Population: Data from one subject not included because subject did not have past positive response to either allergen.
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Groups:
- Disperse Blue 0.017 mg/cm2; Disperse Blue 0.050 mg/cm2; Disperse Blue 0.150 mg/cm2: Concordance between disperse blue and the reference petrolatum allergen
- Bronopol 0.125 mg/cm2; Bronopol 0.250 mg/cm2; Bronopol 0.500 mg/cm2; Bronopol 0.750 mg/cm2: Concordance between bronopol and the reference petrolatum allergen
Arm/Group | Disperse Blue 0.017 mg/cm2 | Disperse Blue 0.050 mg/cm2 | Disperse Blue 0.150 mg/cm2 | Bronopol 0.125 mg/cm2 | Bronopol 0.250 mg/cm2 | Bronopol 0.500 mg/cm2 | Bronopol 0.750 mg/cm2
Number analyzed (Participants) | 21 | 21 | 21 | 26 | 26 | 26 | 26
percentage of agreement | 81.0 [58.1 to 94.6] | 95.2 [76.2 to 99.9] | 90.5 [69.6 to 98.8] | 84.6 [65.1 to 95.6] | 100.0 [86.8 to 100.0] | 76.9 [56.4 to 91.0] | 61.5 [40.6 to 79.8]

7. Secondary Outcome: Frequency of Irritation (Tape Reactions), Late/Persistent Reactions and Subject-reported Itching or Burning
Description: Percentage of subjects who exhibited irritation and itching or burning at patch removal (entire panel is evaluated) and late/persistent reactions.
  Late reactions occur 7-10 days after patch application Persistent reactions initially occur at 2-4 days after application and persist through 7-21 days after application
Time Frame: Day 2-21
Population: Data from one subject not included because subject did not have past positive response to either allergen.
Measure: Number; unit: percentage of participants
Groups:
- Disperse Blue Irritation Reactions: Percentage of subjects who exhibited irritation (tape reactions) to disperse blue panel
- Bronopol Irritation Reactions: Percentage of subjects who exhibited irritation (tape reactions) to bronopol panel
- Disperse Blue Itching and/or Burning: Percentage of subjects who exhibited itching and/or burning to disperse blue panel
- Bronopol Itching and/or Burning: Percentage of subjects who exhibited itching and/or burning to bronopol panel
- Disperse Blue 0.017 Late Reactions; Disperse Blue 0.050 mg/cm2 Late Reactions; Disperse Blue 0.150 mg/cm2 Late Reactions; Negative Control Late Reactions; Bronopol 0.125 mg/cm2 Late Reactions; Bronopol 0.250 mg/cm2 Late Reactions; Bronopol 0.500 mg/cm2 Late Reactions; Bronopol 0.750 mg/cm2 LateReactions: Percentage of subjects who exhibited late reactions
- Disperse Blue 0.017 mg/cm2 Persistent Reactions; Disperse Blue 0.050 mg/cm2 Persistent Reactions; Disperse Blue 0.150 mg/cm2 Persistent Reactions; Negative Control Persistent Reactions; Bronopol 0.125 mg/cm2 Persistent Reactions; Bronopol 0.250 mg/cm2 Persistent Reactions; Bronopol 0.500 mg/cm2 Persistent Reactions; Bronopol 0.750 mg/cm2 Persistent Reactions: Percentage of subjects who exhibited persistent reactions
Arm/Group | Disperse Blue Irritation Reactions | Bronopol Irritation Reactions | Disperse Blue Itching and/or Burning | Bronopol Itching and/or Burning | Disperse Blue 0.017 Late Reactions | Disperse Blue 0.050 mg/cm2 Late Reactions | Disperse Blue 0.150 mg/cm2 Late Reactions | Negative Control Late Reactions | Disperse Blue 0.017 mg/cm2 Persistent Reactions | Disperse Blue 0.050 mg/cm2 Persistent Reactions | Disperse Blue 0.150 mg/cm2 Persistent Reactions | Negative Control Persistent Reactions | Bronopol 0.125 mg/cm2 Late Reactions | Bronopol 0.250 mg/cm2 Late Reactions | Bronopol 0.500 mg/cm2 Late Reactions | Bronopol 0.750 mg/cm2 LateReactions | Bronopol 0.125 mg/cm2 Persistent Reactions | Bronopol 0.250 mg/cm2 Persistent Reactions | Bronopol 0.500 mg/cm2 Persistent Reactions | Bronopol 0.750 mg/cm2 Persistent Reactions
Number analyzed (Participants) | 21 | 26 | 21 | 26 | 21 | 21 | 21 | 21 | 21 | 21 | 21 | 21 | 26 | 26 | 26 | 26 | 26 | 26 | 26 | 26
percentage of participants | 71.4 | 65.4 | 76.2 | 73.1 | 0 | 0 | 0 | 0 | 19.0 | 19.0 | 28.6 | 1.9 | 0 | 0 | 0 | 0 | 11.5 | 15.4 | 11.5 | 11.5

8. Secondary Outcome: Adverse Events
Description: The adverse event-reporting period began at application and ended with the Day 21 visit. Adverse events were followed until they resolved. Serious adverse events and those assessed by the investigator as possibly related to the investigational product were to be followed until they resolved or until the investigator assessed them as chronic or stable.
Time Frame: Days 0-21
Measure: Number; unit: events
Groups:
- Adverse Events Related to Investigational Panel: Number of reported adverse events related to investigational or reference allergens.
- Adverse Events Not Related: Number of adverse events not related to investigational or reference allergens
Arm/Group | Adverse Events Related to Investigational Panel | Adverse Events Not Related
Number analyzed (Participants) | 48 | 48
events | 1 | 1

ADVERSE EVENTS:
Time Frame: Day 1 through Day 21
Description: Serious or possibly related events were to be followed until they resolved or assessed as chronic or stable
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 2/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=48)
Upset stomach (Gastrointestinal disorders) | 1 (1) — Event was not related to the investigational panel.
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — Event could not be attributed to a single allergen or allergen concentration. It was determined to be related to the the entire panel.

LIMITATIONS AND CAVEATS:
There were no limitations or caveats which led to unreadable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No